CLINICAL TRIAL: NCT06798532
Title: Interest of Preoperative Arteriography to Identify the Adamkiewicz Artery Before Surgery for Basi-thoracic Neuroblastic Tumors
Acronym: AKA-NBL
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP241337
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Tumor, Solid; Neuroblastic Tumors; Neuroblastoma
Keywords: Neuroblastic tumors; Neuroblastomas; Ganglioneuroblastomas; Ganglioneuromas; Adamkiewicz Artery; Pediatric surgery
MeSH Terms: conditions — Neoplasms; Neuroblastoma; Ganglioneuroblastoma; Ganglioneuroma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric patients: Patients undergoing surgery for a neuroblastic tumor (neuroblastoma, ganglioneuroblastoma) with basi-thoracic location between T8 and L1, with or without intraspinal component and treated in a pediatric surgery department in France between 2005 and 2024.
  Interventions: Other: Collection of data from the patient's medical file.

INTERVENTIONS:
Other: Collection of data from the patient's medical file. — Collection of data from the patient's medical file.

SUMMARY:
Neuroblastic tumors (NBTs) develop from neural crest cells that give rise to the sympathetic nervous system. They include neuroblastomas, ganglioneuroblastomas, and ganglioneuromas. They represent approximately 10% of solid tumors in children under 15 years of age. In 15 to 20% of cases, NBTs are located in the thoracic region. These paravertebral tumors have an extracanal component and some also have an intraspinal component (dumbbell tumors) that can cause spinal cord compression. Surgery for these tumors also exposes the patient to neurological complications. In the thorax, the basi-thoracic location (T9-T12) may be particularly at risk due to the presence of the artery of Adamkiewicz (AKA), which supplies blood to the spinal cord; damage to this artery can result in spinal cord ischemia. To avoid this scenario, some teams recommend performing spinal cord arteriography to identify AKA. However, many centers do not perform arteriography and do not report more postoperative complications.

Currently, there is no consensus on the indications for performing preoperative spinal arteriography in patients undergoing surgery for basi-thoracic NBT.

This study evaluates the practice in France of preoperative arteriography to identify the AKA among patients undergoing surgery for basi-thoracic neuroblastic tumors and analyzes the incidence of postoperative neurological complications in these patients.

DETAILED DESCRIPTION:
Neuroblastic tumors (NBTs) develop from neural crest cells that give rise to the sympathetic nervous system. They include neuroblastomas, ganglioneuroblastomas, and ganglioneuromas. They represent approximately 10% of solid tumors in children under 15 years of age. In 15 to 20% of cases, NBTs are located in the thoracic region. These paravertebral tumors have an extracanal component and some also have an intraspinal component (dumbbell tumors) that can cause spinal cord compression. Surgery for these tumors also exposes the patient to neurological complications. In the thorax, the basi-thoracic location (T9-T12) may be particularly at risk due to the presence of the artery of Adamkiewicz (AKA), which supplies blood to the spinal cord; damage to this artery can result in spinal cord ischemia. To avoid this scenario, some teams recommend performing spinal cord arteriography to identify AKA. However, many centers do not perform arteriography and do not report more postoperative complications.

Currently, there is no consensus on the indications for performing preoperative spinal arteriography in patients undergoing surgery for basi-thoracic NBT.

This study evaluates the practice in France of preoperative arteriography to identify the AKA among patients undergoing surgery for basi-thoracic neuroblastic tumors and analyzes the incidence of postoperative neurological complications in these patients.

It seems that in France, unlike other European sites, there is no systematic search for the artery of Adamkiewicz before surgery for neuroblastic tumors in most pediatric surgery departments. It does not seem that this is responsible for postoperative neurological complications but this assessment has never been performed.

The hypothesis of the study is that the neurological complications observed postoperatively are due to nerve root surgery or to spinal cord injury by direct trauma through the foramens, but not to spinal cord ischemia.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing surgery for a neuroblastic tumor (neuroblastoma, ganglioneuroblastoma, ganglioneuroma)
2. Basithoracic location between T8 and L1
3. With or without intraspinal component
4. Treated in a pediatric surgery department in France
5. Between 2005 and 2024
6. Adult patients or holders of parental authority of minor patients informed and not opposed to the use of data for the study

Exclusion Criteria:

1. Post-operative follow-up of less than 6 months

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients undergoing surgery for a neuroblastic tumor in a pediatric surgery department in France between 2005 and 2024 and meeting the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of neurological complications secondary to spinal cord ischemia | 2005 to 2024
  Assessment of postoperative neurological complications in patients undergoing surgery for basi-thoracic NBT, with or without preoperative spinal cord arteriography.

SECONDARY OUTCOMES:
Demographic characteristics of patients undergoing surgery for basithoracic neuroblastic tumor | 2005 to 2024
  Describe the demographic characteristics of patients undergoing surgery for basithoracic neuroblastic tumor.
Outcome of patients undergoing surgery for basithoracic neuroblastic tumor | 2005 to 2024
  Describe the overall survival and recurrence-free survival.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna MD Cornet, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Sabine MD, PhD Sarnacki, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (27):
- France (27):
  - CHU d'Amiens, Amiens
  - CHU de Besançon, Besançon
  - CHU de Bordeaux, Bordeaux
  - CHU de Brest, Brest
  - CHU de Lyon, Bron
  - CHU de Caen, Caen
  - CHU de Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - CHU de Lille, Lille
  - CHU de Limoges, Limoges
  - CHU de Marseille, Marseille
  - CHU de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hôpital Trousseau, Paris
  - Hôpital Necker enfants malades, Paris
  - Hôpital Robert Debré, Paris
  - CHU de Poitiers, Poitiers
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de La Réunion, Saint-Denis
  - CHU de Strasbourg, Strasbourg
  - CHU de Toulouse, Toulouse
  - CHU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lindeire S, Hauser JM. Anatomy, Back, Artery of Adamkiewicz. 2025 Mar 25. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK532971/ PMID 30422566
- [Background] Nordin AB, Fallon SC, Jea A, Kim ES. The use of spinal angiography in the management of posterior mediastinal tumors: case series and review of the literature. J Pediatr Surg. 2013 Sep;48(9):1871-7. doi: 10.1016/j.jpedsurg.2013.04.029. PMID 24074660
- [Background] Schmidt A, Hempel JM, Ellerkamp V, Warmann SW, Ernemann U, Fuchs J. The Relevance of Preoperative Identification of the Adamkiewicz Artery in Posterior Mediastinal Pediatric Tumors. Ann Surg Oncol. 2022 Jan;29(1):493-499. doi: 10.1245/s10434-021-10381-8. Epub 2021 Jul 31. PMID 34331163
- [Background] Bosmia AN, Hogan E, Loukas M, Tubbs RS, Cohen-Gadol AA. Blood supply to the human spinal cord: part I. Anatomy and hemodynamics. Clin Anat. 2015 Jan;28(1):52-64. doi: 10.1002/ca.22281. Epub 2013 Jun 27. PMID 23813725
- [Background] De Bernardi B, Gambini C, Haupt R, Granata C, Rizzo A, Conte M, Tonini GP, Bianchi M, Giuliano M, Luksch R, Prete A, Viscardi E, Garaventa A, Sementa AR, Bruzzi P, Angelini P. Retrospective study of childhood ganglioneuroma. J Clin Oncol. 2008 Apr 1;26(10):1710-6. doi: 10.1200/JCO.2006.08.8799. PMID 18375900
- [Background] Furak J, Geczi T, Tiszlavicz L, Lazar G. Postoperative paraplegia after resection of a giant posterior mediastinal tumour. Importance of the blood supply in the upper spinal cord. Interact Cardiovasc Thorac Surg. 2011 May;12(5):855-6. doi: 10.1510/icvts.2010.257105. Epub 2011 Feb 8. PMID 21303870
- [Background] Boglino C, Martins AG, Ciprandi G, Sousinha M, Inserra A. Spinal cord vascular injuries following surgery of advanced thoracic neuroblastoma: an unusual catastrophic complication. Med Pediatr Oncol. 1999 May;32(5):349-52. doi: 10.1002/(sici)1096-911x(199905)32:53.0.co;2-p. PMID 10219336